CLINICAL TRIAL: NCT02494310
Title: Point-of-Care, Real-Time Optical Imaging to Enable Screening for Cervical Cancer and Its Precursors in Low-Resource Settings
Brief Title: HRME: Screening for Cervical Cancer and Its Precursors in Low-Resource Settings
Acronym: HRME-UH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: William Marsh Rice University (Other); M.D. Anderson Cancer Center (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jose Humberto Tavares Guerreiro Fregnani, PhD, Barretos Cancer Hospital, Barretos Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HRME-UH2
Record Dates: First submitted 2015-07-06; First posted 2015-07-10 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Neoplasia of the Uterine Cervix; Cancer Prevention; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HRME - Prevention Mobile Unit (Experimental): Procedures to be done in the mobile unit (van): Visual inspection will be performed with 5% acetic acid (VIA) applied to the cervix followed by standard colposcopy. Proflavine (0.01%) will then be applied topically. Lugol's solution will then be applied and colposcopy performed and abnormal lesions noted. HRME images will be acquired from any areas that are abnormal by VIA and/or colposcopy. VIA, colposcopy and HRME observations will recorded by quadrant. Any abnormal areas by VIA and/or colposcopy will be biopsied. If no abnormal areas are noted, one cervical biopsy will be obtained from a normal appearing area with a HRME image of this area obtained.
  Interventions: Device: High-Resolution Microendoscopy Imaging
- HRME - Barretos Cancer Hospital (Experimental): Procedures to be done at Barretos Cancer Hospital: Visual inspection will be performed with 5% acetic acid (VIA) applied to the cervix followed by standard colposcopy. Proflavine (0.01%) will then be applied topically. Lugol's solution will then be applied and colposcopy performed and abnormal lesions noted. HRME images will be acquired from any areas that are abnormal by VIA and/or colposcopy. VIA, colposcopy and HRME observations will recorded by quadrant. Any abnormal areas by VIA and/or colposcopy will be biopsied. If no abnormal areas are noted, one cervical biopsy will be obtained from a normal appearing area with a HRME image of this area obtained.
  Interventions: Device: High-Resolution Microendoscopy Imaging

INTERVENTIONS:
Device: High-Resolution Microendoscopy Imaging — Innovative technique to evaluate epithelial cell morphology in situ. The device is not invasive and does not exchange energy with human body.
  Other Names: HRME

SUMMARY:
A new mobile diagnostic and treatment unit is being developed by BCH to address the loss-to follow-up associated with the mobile screening program and demonstrate POC diagnosis by HRME. The mobile diagnostic and treatment unit will be equipped with the tools and infrastructure necessary to perform HRME, VIA, colposcopy, biopsy and treatment with cryotherapy. A team of a colposcopist, nurse, nursing assistant, and driver will staff the mobile diagnostic and treatment unit. The unit will travel to offer follow-up diagnostic and treatment services to women who have screened positive during a prior visit with the mobile screening unit. The mobile diagnostic and treatment unit will be constructed and maintained at BCH.

DETAILED DESCRIPTION:
A new mobile diagnostic and treatment unit is being developed by BCH to address the loss-to follow-up associated with the mobile screening program and demonstrate POC diagnosis by HRME. The mobile diagnostic and treatment unit will be equipped with the tools and infrastructure necessary to perform HRME, VIA, colposcopy, biopsy and treatment with cryotherapy. A team of a colposcopist, nurse, nursing assistant, and driver will staff the mobile diagnostic and treatment unit. The unit will travel to offer follow-up diagnostic and treatment services to women who have screened positive during a prior visit with the mobile screening unit. The mobile diagnostic and treatment unit will be constructed and maintained at BCH.

The study will include 200 women with abnormal Pap tests identified through BCH's existing mobile screening program. Participants will be randomized by cluster to receive follow up care either through the new mobile diagnostic and treatment unit (experimental arm) or through recall to BCH (standard of care). We are using cluster randomization to avoid contamination between arms because some women getting mobile unit services may be concerned that they are getting lesser services than what they could get at BCH or some women being referred to BCH may resent not having the convenience of a mobile unit. Because the areas visited by the mobile units are geographically isolated, we do not anticipate any patients crossing over to the other study arm.

VIA will be performed with 5% acetic acid applied to the cervix and any abnormal lesions noted. Standard colposcopy will then be performed and abnormal lesions noted. Proflavine (0.01%) will then be applied topically. Lugol's solution will then be applied and colposcopy performed and abnormal lesions noted. Proflavine (0.01% will then be reapplied. HRME images will be acquired from any areas that are abnormal by VIA and/or colposcopy. In addition, all 4 quadrants will be probed by HRME (4Q HRME) to ensure that non-acetowhite lesions are also located. The provider will note their impression of the lesion and the HRME image at each site (normal, benign, low-grade precancer, high grade precancer or cancer). The entire HRME imaging procedure should add less than 10 minutes to the standard colposcopy exam. VIA, colposcopy and HRME observations will recorded by quadrant. Any abnormal areas by VIA and/or colposcopy will be biopsied. If no abnormal areas are noted, one cervical biopsy will be obtained from a normal appearing area with a HRME image of this area obtained. Two expert pathologists, blinded to all study results, will review histology and classify as either normal, CIN1, CIN2, CIN3, AIS or cancer, according to standard criteria; discrepant results will be resolved by consensus review.

TREATMENT:

Women randomized to the mobile diagnostic and treatment unit who have a HSIL Pap and/or a lesion noted by VIA and/or colposcopy will undergo immediate treatment with cryotherapy following biopsies, provided the lesion meets the following criteria: 1) covers <75% of the ectocervix; 2) can be fully covered with the cryotherapy tip; 3) does not extend into the endocervical canal. If the colposcopic findings are concerning for invasive cancer or the lesion is not amenable to treatment with cryotherapy, the patient will be referred immediately to BCH for additional evaluation and treatment per standard of care.

Women with a biopsy showing CIN2+ who did not undergo cryotherapy due to a negative VIA/colposcopy, will be recalled to BCH immediately for LEEP (CIN2/3). Women with a biopsy showing CIN2/3 who underwent cryotherapy will be recalled to BCH or the mobile unit for a 6-month follow-up visit. If persistent or recurrent disease is noted, they will be referred to BCH for further treatment. Women with a biopsy showing cancer of adenocarcinoma in situ (AIS) will be recalled to BCH immediately for cold knife cone (CKC) or other evaluation and treatment per standard of care regardless of whether or not cryotherapy was performed. Women with CIN1 or less will return for follow-up to the mobile unit or BCH for follow-up at 12 months. Women randomized to return to a central facility for follow up care will undergo VIA, colposcopy, HRME and biopsies as described above. Patients found to have CIN2+ will be treated per standard of care at BCH.

ELIGIBILITY:
Inclusion Criteria:

1. Women with an abnormal Pap test (atypical squamous cells of undetermined significance or more severe interpretations [≥ASC-US])
2. Women with an intact cervix (patients who have undergone previous LEEP, cone and/or cryotherapy are eligible)
3. Women of childbearing potential must have a negative urine or serum pregnancy test
4. Women who are at least 18 years of age or older
5. Ability to understand and the willingness to provide informed consent and sign a written Informed Consent Document (ICD)

Exclusion Criteria:

1. Women <18 years of age
2. Women who have undergone a hysterectomy with removal of the cervix
3. Women with a known allergy to proflavine or acriflavine
4. Women who are pregnant or nursing
5. Women unable or unwilling to provide informed consent or sign a written Informed Consent Document (ICD)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment completion rate. | Participants will be followed for two years.
  Treatment completion for screen-positive women invited to visit a mobile diagnostic and treatment unit in their local area compared to those who are asked to return to a central facility for diagnosis and treatment.

SECONDARY OUTCOMES:
Efficacy (ability to detect CIN 2+ in women with previous abnormal Pap test). | 6 months
  Efficacy of HRME in detecting CIN 2+ in women with previous abnormal Pap test.